CLINICAL TRIAL: NCT06472726
Title: Mental Health App for Cancer Survivors Study
Acronym: MACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: App developer is no longer in business
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0111; 5P50CA278595-07 (NIH); UW23133 (Other: UW Madison); A532007 (Other: UW Madison); SMPH/FAMILY MED/RES GRANTS (Other: UW Madison); Protocol version 2/10/2025 (Other: UW Madison)
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer; Head and Neck Cancers; Depression
MeSH Terms: conditions — Head and Neck Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IONA Mind app (Experimental): Participants will be asked to use the IONA Mind app for a 6-week period.
  Interventions: Behavioral: IONA Mind app

INTERVENTIONS:
Behavioral: IONA Mind app — The IONA Mind app is a smartphone app that delivers mental health support.

SUMMARY:
The goal of this clinical trial is to adapt a mental health digital app to treat depression among head and neck cancer patients and survivors.

Participants will download and use the digital mental health app for a 6-week period, and will complete related surveys.

DETAILED DESCRIPTION:
This study is being done to estimate the feasibility/efficacy/acceptability of the IONA Mind app for head and neck cancer (HNC) patients and survivors who show evidence of comorbid depression.

IONA Mind is a digital app that delivers mental health support. Once users sign up and respond to the initial assessment with PHQ-9 questionnaire, it reaches out to users proactively to offer support, personalized wellbeing plans, and guidance.

In partnership with the UWCCC, the IONA Mind Team, the Survey of the Health of Wisconsin (SHOW) and the Head Neck Patient Advocacy team, the investigators propose adaptation of the IONA Mind app and pilot testing the app with 30 HNC patients and survivors. Using a mixed method design the specific aims are:

* AIM 1. Adaptation of IONA Mind app for head and neck cancer. The research team will iteratively adapt the IONA Mind app to provide psychological support for HNC patients and survivors. The HNC Survivors Advisory Board will assist in identifying key aspects of the HNC survivors' journey from diagnosis to the survivorship phase, which will be prioritized and considered to iteratively redesign the IONA Mind phone app to better support HNC patients and survivors
* AIM 2. Identify feasibility of the IONA Mind app for head and neck cancer. The IONA Mind app will be tested with 30 HNC patients and survivors, recruited from the Survey of the Health of Wisconsin (SHOW) recruitment registry and from the clinical practice at UW Carbone Cancer Center (UWCCC)
* AIM 3. Determine preliminary efficacy IONA Mind app tailored for depression comorbid with head and neck cancer. Clinical outcomes will be measured at baseline, weekly for 6 weeks (including the 6-week period of app utilization), and post-intervention follow-up conducted at 1- and 3-month post intervention using validated tools to access depression
* AIM 4. Determine satisfaction and acceptability of the IONA Mind app. Satisfaction with the IONA Mind app will be measured with the System Usability Scale (SUS) delivered at 1-2 weeks following the completion of the app utilization. In addition, a qualitative interview for a random sub sample of 10 - 15 participants will occur shortly after completion of the intervention to assess satisfaction with and acceptability of the mobile app. A head and neck patient and survivor phone app Low-Intensity Cognitive Behavioral Therapy (LiCBT) intervention to treat depression co-designed by HNC advocates, mental health professionals and an expert technologist is a critical outcome of this research.

ELIGIBILITY:
Inclusion Criteria:

* History of HNC confirmed by histopathologic diagnosis. The signed report must be available on electronic health record (EHR) for participants who received treatment or follow-up at University of Wisconsin Carbone Cancer Center (UWCCC). Alternatively, participants must have a printed signed report if received treatment out of UWCCC
* Age greater than or equal to 22 years at the time of consent
* Patient Health Questionnaire-9 (PHQ-9) score ≥ 5 and ≤ 19 (moderate and severely moderate depression)
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Unable to read and speak English.
* Utilization of prescription medicine for depression.
* Patient Health Questionnaire-9 (PHQ-9) score of greater than or equal to 20 (severe depression)
* Patient Health Questionnaire-9 (PHQ-9) score greater than or equal to 1 on the suicidal question (question 9)
* Pregnant people

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Feasibility: Screening to enrollment ratio | baseline
  Recruitment and Retention Tracking Tool will calculate the screening to enrollment ratio.
Feasibility: Measured by Retention rate | up to 20 weeks
  The Recruitment and Retention Tracking Tool will calculate the the number of participants who are recruited, dropped out, and complete the intervention.
Feasibility: IONA Mind app Utilization in Minutes | up to 20 weeks
  Minutes of app usage
Change in Patient Health Questionnaire-9 (PHQ-9) | baseline, weekly during intervention from weeks 1 through 6, 1-month post intervention, 3-month post intervention (up to 20 weeks in total)
  Clinical outcomes will be measured at baseline, weekly for 6 weeks during app utilization, and at post-intervention follow-up conducted at 1- and 3-month post intervention using the PHQ-9. The PHQ-9 is a 9-item scale assessing depression. It is scored on a 0- to 3-point Likert scale where 0=Not at all and 3 = nearly every day. Mean scores are reported for a range from 0-27 where higher scores indicate greater levels of depression
Satisfaction Measured by System Usability Scale | 2 weeks post-intervention (up to 8 weeks on study)
  The System Usability Scale is a 10-item questionnaire assessing participants' satisfaction with the IONA Mind app. It is scored on a 1- to5-point Likert scale where 1= strongly disagree and 5= strongly agree. Mean item scores are reported with a range from 10 to 50 where higher scores indicate greater satisfaction with the app.
Qualitative Measure of Acceptability | 2 weeks post-intervention (up to 8 weeks on study)
  Ascertained via a qualitative semi-structured interview for a random subsample of 10 - 15 participants after completion of the intervention (1-2 weeks post-intervention). Interview answers with be coded for thematic analysis and reported by participant count.

CONTACTS AND LOCATIONS:
Overall Officials: Earlise Ward, MS, PhD, LP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No